CLINICAL TRIAL: NCT03465982
Title: Timing to Minimally Invasive Surgery After Neoadjuvant Chemoradiotherapy for Rectal Cancer: a Multicenter Randomised Controlled Trial
Brief Title: Timing to Minimally Invasive Surgery After Neoadjuvant Chemoradiotherapy for Rectal Cancer
Acronym: TiMiSNAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Responsible Party: Principal Investigator, Igor Monsellato, Principal Investigator, Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1/18
Record Dates: First submitted 2018-02-23; First posted 2018-03-15 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; robotic rectal cancer resection; minimally invasive surgery; Colorectal Cancer; chemoradiation treatment rectal cancer
MeSH Terms: conditions — Rectal Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Interval Time Arm (Active Comparator): Minimally invasive surgery after 8 weeks from chemoradiation treatment
  Interventions: Procedure: Surgery after 8 weeks from chemoradiation treatment
- Delayed Interval Time Arm (Active Comparator): Minimally invasive surgery after 12 weeks from chemoradiation treatment
  Interventions: Procedure: Surgery after 12 weeks from chemoradiation treatment

INTERVENTIONS:
Procedure: Surgery after 8 weeks from chemoradiation treatment — Minimally invasive surgery after 8 weeks from chemoradiation treatment
  Arms: Standard Interval Time Arm
Procedure: Surgery after 12 weeks from chemoradiation treatment — Minimally invasive surgery after 12 weeks from chemoradiation treatment
  Arms: Delayed Interval Time Arm

SUMMARY:
The trial is a multicenter, prospective, randomized controlled, unblinded, parallel-group trial comparing standard and delayed surgery after neoadjuvant chemoradiotherapy for the curative treatment of rectal cancer. Three-hundred and thirty-two patients will be randomized on an equal basis to either robotic-assisted/standard laparoscopic rectal cancer surgery after 8 weeks or robotic-assisted/standard laparoscopic rectal cancer surgery after 12 weeks. The recruiting interval will be of 5 years and the follow-up period will end 5 years after the last patient is randomized.

DETAILED DESCRIPTION:
PURPOSE

To demonstrate if delayed timing of surgery after neoadjuvant chemoradiotherapy actually affects pathological complete response (pCR) and reflects on disease-free survival (DFS) and overall survival (OS) rather than standard timing. Eight weeks are the current standard interval to surgery after neoadjuvant treatment, while 12 weeks represent the "minimum" longer time interval to determine further tumor modifications and the "a priori" choice to avoid hypothetical surgical detrimental effect (postoperative complications related to radiation therapy).

Primary Endpoint

* pCR

Secondary Endpoints

* DFS
* OS
* QoL (quality of Life)

Site Eligibility

The trial is a multicenter collaboration, involving all those centers able to provide the standard of cure for locally advanced rectal cancer. All the involved centers have to respect the following criteria:

* Site able to perform robotic-assisted and standard laparoscopic rectal cancer surgery and TaTME (transanal total mesorectal excision)
* Site able to provide a preoperative work up according to the work up criteria specified in this trial
* Site able to provide standard neoadjuvant treatment, both chemo and radiation therapy, according to the criteria specified in this trial
* Predicted capability to recruit a minimum of 15 patients per year to the trial.

Randomization will take place after consent is obtained and after patients have completed their baseline patient reported questionnaires. Patient consent and randomization will take place as close to the date of start of the neoadjuvant treatment as possible and must be no more than 30 days prior to planned treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* cT3/4N0/+M0 confirmed on CT-scan, MRI (stratification for T3a-b-c-d) 3
* Tumor starting from the distal or medium rectum (even those crossing the peritoneal reflection at distal margin, within 15 cm from the anal margin)
* Histologically-proven adenocarcinoma of the rectum
* Eligible for a resective surgery with TME (low anterior resection, intersphincteric resection, abdominoperineal resection)
* Eligible for resection by minimally-invasive surgery (standard or robotic-assisted laparoscopic procedure, all robotic systems will be accepted)
* Eligible for chemoradiation treatment
* Able to give written informed consent
* Capable of completing required questionnaires at time of consent (provided questionnaires are available in a language spoke fluently by the participant)

Exclusion Criteria:

* Metastatic disease
* Squamous carcinoma of the anal canal
* Synchronous colorectal tumors requiring multi-segment surgical resection (n.b. a benign lesion within the resection field in addition to the main cancer would not exclude a patient)
* History of psychiatric or addictive disorder or other medical condition that, in the opinion of the investigator, would preclude the patient from meeting the trial requirements
* Pregnancy
* Unable to complete neoadjuvant treatment
* Unable to give free informed consent
* Previous radiation treatment on the pelvis
* Inflammatory bowel disease
* Hereditary colorectal disease
* Previous tumors other than non-melanoma skin cancer, papillary or follicular thyroid cancer
* Participation in another rectal cancer clinical trial relating to the topic of this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2018-06-05 (Actual); Primary Completion 2025-06-05 (Estimated); Study Completion 2029-06-05 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response (pCR) | 8-12 weeks
  Pathologic Complete response on cancer defined as absence of cancer cells on specimen

SECONDARY OUTCOMES:
DFS | 5 years
  Disease Free survival
OS | 5 years
  Overall Survival

CONTACTS AND LOCATIONS:
Locations (14):
- Italy (14):
  - SS. Antonio e Biagio e Cesare Arrigo Hospital, Alessandria, AL
  - Ospedale Gian Battista Morgagni - Luigi Pierantoni, Forlì, Forlì-Cesena
  - Ospedale Civile Pietro Cosma, Camposampiero, Padua
  - Ospedale Sacro Cuore, Negrar, Verona
  - Ente Ecclesiastico ospedale generale Regionale Miulli, Acquaviva delle Fonti
  - Ospedale degli Infermi, Biella
  - Istituto del Radio Olindo Alberti, Spedali Civili di Brescia, Brescia
  - ASST Ospedale di Cremona, Cremona
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Ospedale Maggiore Policlinico Fondazione Ca' Granda, Milan
  - Ospedale San Raffaele IRCCS, Milan
  - Istituto Nazionale Tumori - IRCCS Fondazione G. Pascale, Napoli
  - Ospedale San Francesco, Nuoro
  - Azienda Ospedaliera San Giovanni - Addolorata, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sauer R, Becker H, Hohenberger W, Rodel C, Wittekind C, Fietkau R, Martus P, Tschmelitsch J, Hager E, Hess CF, Karstens JH, Liersch T, Schmidberger H, Raab R; German Rectal Cancer Study Group. Preoperative versus postoperative chemoradiotherapy for rectal cancer. N Engl J Med. 2004 Oct 21;351(17):1731-40. doi: 10.1056/NEJMoa040694. PMID 15496622
- [Result] Petrelli F, Sgroi G, Sarti E, Barni S. Increasing the Interval Between Neoadjuvant Chemoradiotherapy and Surgery in Rectal Cancer: A Meta-analysis of Published Studies. Ann Surg. 2016 Mar;263(3):458-64. doi: 10.1097/SLA.0000000000000368. PMID 24263329
- [Result] Erlandsson J, Holm T, Pettersson D, Berglund A, Cedermark B, Radu C, Johansson H, Machado M, Hjern F, Hallbook O, Syk I, Glimelius B, Martling A. Optimal fractionation of preoperative radiotherapy and timing to surgery for rectal cancer (Stockholm III): a multicentre, randomised, non-blinded, phase 3, non-inferiority trial. Lancet Oncol. 2017 Mar;18(3):336-346. doi: 10.1016/S1470-2045(17)30086-4. Epub 2017 Feb 10. PMID 28190762
- [Result] Kaytan-Saglam E, Balik E, Saglam S, Akgun Z, Ibis K, Keskin M, Dagoglu N, Kapran Y, Gulluoglu M. Delayed versus immediate surgery following short-course neoadjuvant radiotherapy in resectable (T3N0/N+) rectal cancer. J Cancer Res Clin Oncol. 2017 Aug;143(8):1597-1603. doi: 10.1007/s00432-017-2406-6. Epub 2017 Apr 3. PMID 28374169
- [Result] Lefevre JH, Mineur L, Kotti S, Rullier E, Rouanet P, de Chaisemartin C, Meunier B, Mehrdad J, Cotte E, Desrame J, Karoui M, Benoist S, Kirzin S, Berger A, Panis Y, Piessen G, Saudemont A, Prudhomme M, Peschaud F, Dubois A, Loriau J, Tuech JJ, Meurette G, Lupinacci R, Goasgen N, Parc Y, Simon T, Tiret E. Effect of Interval (7 or 11 weeks) Between Neoadjuvant Radiochemotherapy and Surgery on Complete Pathologic Response in Rectal Cancer: A Multicenter, Randomized, Controlled Trial (GRECCAR-6). J Clin Oncol. 2016 Nov 1;34(31):3773-3780. doi: 10.1200/JCO.2016.67.6049. PMID 27432930
- [Derived] Monsellato I, Alongi F, Bertocchi E, Gori S, Ruffo G, Cassinotti E, Baldari L, Boni L, Pernazza G, Pulighe F, De Nisco C, Perinotti R, Morpurgo E, Contardo T, Mammano E, Elmore U, Delpini R, Rosati R, Perna F, Coratti A, Menegatti B, Gentilli S, Baroffio P, Buccianti P, Balestri R, Ceccarelli C, Torri V, Cavaliere D, Solaini L, Ercolani G, Traverso E, Fusco V, Rossi M, Priora F, Numico G, Franzone P, Orecchia S. Standard (8 weeks) vs long (12 weeks) timing to minimally-invasive surgery after NeoAdjuvant Chemoradiotherapy for rectal cancer: a multicenter randomized controlled parallel group trial (TiMiSNAR). BMC Cancer. 2019 Dec 16;19(1):1215. doi: 10.1186/s12885-019-6271-3. PMID 31842784

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-28): https://cdn.clinicaltrials.gov/large-docs/82/NCT03465982/Prot_SAP_005.pdf